CLINICAL TRIAL: NCT00027079
Title: Combined Pharmacotherapies for Alcoholism (Naltrexone/Ondansetron)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAJOH12964
Record Dates: First submitted 2001-11-20; First posted 2001-11-21 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Naltrexone; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: ondansetron (Zofran)
Drug: naltrexone (ReVia)
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
This study will compare the effectiveness of ondansetron (Zofran) and naltrexone (ReVia) both alone and in combination in treating Early Onset Alcoholics versus Late Onset Alcoholics. All subjects will received standardized Cognitive Behavioral Therapy. Followup assessments will be completed at 1, 3, 6, and 9 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of alcohol dependence.
* Provide a written informed consent.
* Must weigh within 30% of their ideal body weight.
* Patients must weigh at least 89 lbs. and no more than 342 lbs.
* Good physical health.
* Currently drinking 14 or more alcohol units per week for women and 21 or more alcohol units per week for men in the last 30 days.
* Provide evidence of stable residence in the last month prior to enrollment in the study.
* No plans to move in the nine months after entering the study.
* Literate in English and able to read, understand, and complete questionnaires and follow instructions.
* Willingness to participate in behavioral treatment for alcoholism.

Exclusion Criteria:

* Current psychiatric disorder other than alcohol or nicotine dependence.
* Elevated liver enzymes or elevated bilirubin.
* Severe alcohol withdrawal symptoms which require treatment.
* Serious medical co-morbidity requiring medical intervention or close supervision.
* Severe or life-threatening adverse reactions to medications in the past or during this trial.
* Female patients who are pregnant, lactating, or not adhering to an acceptable form of contraception at any time during the study.
* Received inpatient or outpatient treatment for alcohol dependence within the last 30 days.
* Compelled to participate in an alcohol treatment program for alcohol dependence to maintain their liberty.
* Members of the same household.
* Tuberculosis.
* Current treatment with any medications having a potential effect on alcohol consumption and related behaviors or mood.
* Urine must be free of opiates, cocaine, amphetamines, barbiturates, benzodiazepines, prescription and non-prescription drugs.
* Pyrexia of unknown origin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2001-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States